CLINICAL TRIAL: NCT02113566
Title: A Double-Blind, Repeat-Dose, Parallel Group Study Comparing the Efficacy and Safety of Orally Administered Ibuprofen and Placebo in Delayed Onset Muscle Soreness.
Brief Title: A Study Comparing the Efficacy and Safety of Orally Administered Ibuprofen and Placebo in Delayed Onset Muscle Soreness
Acronym: DOMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jean Brown Research (Other)
Responsible Party: Principal Investigator, Derek Muse, Derek Muse, MD, Jean Brown Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JBR-001
Record Dates: First submitted 2014-04-06; First posted 2014-04-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: Delayed onset muscle soreness; DOMS
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 2 capsules identical to comparator, 3 times daily on Day 1 and Day 2. On Day 3 only one dose will be taken. The intervention is Acetaminophen 1000mg.
  Interventions: Drug: Acetaminophen 1000mg
- Ibuprofen (Active Comparator): 2oomg capsules (400 mg per dose), 3 times daily on Day 1 and Day 2. On Day 3 only one dose will be taken. The intervention is Acetaminophen 1000mg.
  Interventions: Drug: Acetaminophen 1000mg

INTERVENTIONS:
Drug: Acetaminophen 1000mg — Subjects who require rescue medication between hours 4 and 6 will be allowed to take Dose 2 of the study medication. If the subject chooses to take a rescue analgesic (acetaminophen 1000mg), they will be considered a treatment failure. This intervention will be use for the placebo and Ibuprofen arm.
  Other Names: Tylenol

SUMMARY:
The hypotheses to be tested are: Efficacy: Ibuprofen will be more effective than the Placebo in relieving muscle pain/soreness over 48 hour post-dosing with study medication. Safety: There will be no or minimal increased incidence of adverse events (AEs) with Ibuprofen versus and both will be well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* are male or female, 18-55 years of age
* are a sexually active female of childbearing potential willing to use a medically acceptable form of birth control throughout the study and for 30 days following the end of study participation
* have a history of experiencing muscle soreness after moderately strenuous exercise
* are in good general health, with a BMI less than or equal to 30, and able to perform the exercise regimen
* are able to read, comprehend, and sign the informed consent form
* develop muscle pain/soreness within 24-48 hours of the end of the exercise regimen and have a baseline muscle pain/soreness with movement of greater than or equal to 5 on the NRS (numerical rating scale) and at least "moderate" on the categorical scale

Exclusion Criteria:

* regularly works out or exercises the upper extremities with weights or gym equipment during the past 6 months
* works in an occupation that requires regular heavy lifting or involvement of the upper extremities (eg: mover, construction workers)
* allergy or intolerance to any non-steroidal anti-inflammatory drug (NSAID), aspirin or acetaminophen
* the presence of any medical condition (eg: history of bleeding ulcers or current peptic ulcer disease) that would preclude the subject from safely participating in the study'
* any form of arthritis that requires prescription or over-the-counter (OTC)treatment pregnant or lactating female
* current habituation or history of chronic use of analgesic or drugs or severe chronic pain problems that do not respond to OTC medication and/or requires a prescription analgesic
* currently on chronic NSAID therapy for any reason
* current or recent history of drug or alcohol abuse
* has taken an analgesic medication within 5 half lives of performing the exercise regimen during the run-in period or completing the baseline assessment
* has donated blood within the past 30 days
* is unable to swallow whole or large tablets or capsules
* is unable/unwilling to remain at the study center for the 6 hour inpatient observation period.
* participation in an investigational study within the past 30 days of screening
* prior participation in this trial
* site employee or close relative of a site employee directly involved in the conduct or the study or is an employee or close relative of the study doctor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
SPID (Sum Pain Intensity Difference) | 0-48 hours
  The primary efficacy parameter is muscle pain/soreness with movement at 48 hours (SPID 0-48)

SECONDARY OUTCOMES:
spontaneous muscle pain/soreness | 0-48 hours
Muscle stiffness with movement | 0-48 hours
Overall evaluation measures | 0-48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Derek Muse, MD, Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States